CLINICAL TRIAL: NCT07345767
Title: Hypknowledge Nationwide Sleep Extension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Associate Professor of Psychiatry, University of Arizona
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008934275
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Short Sleep Duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group receives standard feedback, where they will be asked to maintain a consistent sleep schedule irrespective of what the Fitbit data or sleep diary report.
- Intervention: Sleep Diary (Experimental): This arm receives weekly feedback on their sleep schedule based on sleep diary data.
  Interventions: Behavioral: Sleep Diary
- Intervention: Fitbit (Experimental): This arm receives weekly feedback on their sleep schedule based on Fitbit data.
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: Sleep Diary — Based on the participant's sleep diary data, a new weekly sleep schedule will be prescribed as follows: if sleep efficiency is <85%, the prescribed time in bed is reduced by 15 minutes (reducing sleep opportunity by 15 minutes); if sleep efficiency is 85-90%, the schedule remains unchanged; if sleep efficiency is >90%, the prescribed time in bed is increased by 15 minutes, allowing an extra 15 minutes of sleep opportunity.
  Arms: Intervention: Sleep Diary
Behavioral: Fitbit — Based on the participant's Fitbit data, a new weekly sleep schedule will be prescribed as follows: if sleep efficiency is <85%, the prescribed time in bed is reduced by 15 minutes (reducing sleep opportunity by 15 minutes); if sleep efficiency is 85-90%, the schedule remains unchanged; if sleep efficiency is >90%, the prescribed time in bed is increased by 15 minutes, allowing an extra 15 minutes of sleep opportunity.
  Arms: Intervention: Fitbit

SUMMARY:
The main goal of this study is to evaluate whether a manually determined sleep extension intervention is effective at improving sleep and related outcomes among adults who find it difficult to get enough sleep.

DETAILED DESCRIPTION:
Approximately 1/3 of Americans sleep ≤6h per night, an amount that has been deemed sub-optimal by the American Academy of Sleep Medicine and Sleep Research Society, the National Sleep Foundation, American Thoracic Society, and the American Heart Association. These consensus statements echo findings from many reviews on this topic. This is alarming, given epidemiologic and experimental research showing that reduced sleep time is associated with a variety of negative health outcomes including obesity, diabetes, cardiovascular disease, and mortality. Different people may need different amounts of sleep and some people may not be able to make large changes to their sleep schedule all at once. Many individuals have situational constraints that change over time. As such, short sleep represents an unmet public health problem. There are, however, no empirically supported interventions for insufficient sleep. The proposed study addresses this critical gap by evaluating the efficacy of a novel intervention that is theoretically grounded, feasible, and has positive impacts on sleep duration. The intervention in the proposed study is by design self-correcting, individually-tailored, and not dependent on unknown individual sleep needs. It can adapt to any schedule and situation and can adapt to changes in a person's sleep schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18-60 years old
2. Have a typical sleep schedule of <=6 hours per night
3. Must have a FitBit device (any model) with Heart Rate Monitor
4. Must have bedtime between 8 pm and 1 am
5. Must have a waketime between 5 am and 10 am
6. Must not have insomnia as determined by diagnosis or score on the Insomnia Severity Index (ISI), or must be treated.
7. Must not have sleep apnea as determined by diagnosis or STOP-BANG scale, or must be treated.
8. Must have a computer or smartphone device for daily sleep diaries.
9. Must have an initial sleep efficiency of at least 85% as determined by sleep diaries and actigraphy.

Exclusion Criteria:

1. Any condition that the PI considers would significantly impede participation in the study.
2. Participant is under 18 years of age or older than 60 years of age
3. Does not own a FitBit device with Heart Rate Monitor
4. Sleep >6 hours per night.
5. Typical bedtime before 8 pm or after 1 am
6. Typical waketime before 5 am or after 10 am
7. Diagnosed with sleep disorders including insomnia or sleep apnea
8. Diagnosed mental health disorder which may impact sleep (i.e. Bipolar Disorder)
9. Taking medications that may affect sleep.
10. Baseline sleep efficiency less than 85%.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1038 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Duration | 9 weeks from enrollment to the end of the study
  Measured in minutes. It is trended from enrollment until the end of the study

SECONDARY OUTCOMES:
Mental Health | 9 weeks from enrollment to the end of the study
  Assessed pre and post-study using questionnaires
Sleepiness/Fatigue | 9 weeks from enrollment to end of the study
  Assessed pre and post-study using questionnaires
Cognitive Functioning | 9 weeks from enrollment to the end of the study
  Assessed pre and post-study using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Grandner, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States